CLINICAL TRIAL: NCT02073058
Title: Evaluation of the Accuracy of the Abbott Sensor Based Interstitial Glucose Monitoring System
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-13128
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Subjects with Type 1 or Type 2 Diabetes Requiring Multiple daily Insulin Injection (MDI) or Continuous Subcutaneous Insulin Infusion (CSII)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: No treatment

SUMMARY:
The purpose of this study is to demonstrate point accuracy of the Abbott Sensor Based Glucose Monitoring (GM) System interstitial glucose results against Reader capillary Blood Glucose (BG) reference using the Consensus Error Grid. During the course of the wear duration, the subject is required to test fingerstick glucose measurement at least eight (8) times a day for capillary reference glucose measurements and three in-clinic visits of a maximum 13 hours each for venous reference glucose measurements. With every reference measurement, the subject or study staff will perform a measurement on the System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must have type 1 or type 2 diabetes for at least 2 years prior to enrollment.
3. Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily) for at least 6 months prior to enrollment.
4. Subject must be able to read and understand English.
5. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
6. Subject must be available to participate in all study visits.
7. Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

1. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
2. Subject is pregnant, attempting to conceive or not willing and able to practice birth control during the study duration (applicable to female subjects only).
3. Subject has skin lesions, scarring, redness, infection or edema at the application sites that could interfere with device placement or the accuracy of interstitial glucose measurements.
4. Subject currently is participating in another clinical trial.
5. Subject has donated blood within 112 days (3.7 months) prior to the beginning of the study activities.
6. Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff. Such conditions include but are not limited to:

   • History of HIV, Hepatitis B or C
7. Subject has a known medical condition that, in the opinion of the investigator, may increase the risk of bleeding.
8. Subject has X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
9. Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 1 or type 2 diabetes who require multiple daily insulin injections (MDI) or continuous subcutaneous insulin infusion (CSII). No more than 20 subjects will have HbA1c > 8.5%, and no more than 20 subjects will have HbA1c < 7% based on the subject screening.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Clinical point accuracy as assessed by the Consensus Error Grid | 14 days

SECONDARY OUTCOMES:
Safety endpoints that include signs and symptoms related to sensor application site | 14 days
Composite measure: Technical point accuracy (difference measures, Bland-Altman analysis, regression and percentage within ranges of the reference) | 14 days
Composite measure: Clinical point accuracy (Clarke Error Grid), trend accuracy (R-deviation, Rate Error Grid and Continuous Glucose Error Grid) and lag time, performance of notifications (sensitivity and false notifications) and questionnaire responses. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute; Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates; Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research; Leslie Klaff, MD, Principal Investigator — Rainier Clinical Research
Locations (4):
- United States (4):
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rainier Clinical Research Center, Renton, Washington

REFERENCES:
- [Derived] Bailey T, Bode BW, Christiansen MP, Klaff LJ, Alva S. The Performance and Usability of a Factory-Calibrated Flash Glucose Monitoring System. Diabetes Technol Ther. 2015 Nov;17(11):787-94. doi: 10.1089/dia.2014.0378. Epub 2015 Jul 14. PMID 26171659